CLINICAL TRIAL: NCT02076204
Title: Mother and Infant Home Visiting Program Evaluation (MIHOPE) - Strong Start
Brief Title: Mother and Infant Home Visiting Program Evaluation-Strong Start
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MDRC (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency); Mathematica Policy Research, Inc. (Other); Johns Hopkins University (Other); James Bell Associates (Unknown); Office of Planning, Research & Evaluation (U.S. Federal Agency)
Responsible Party: Principal Investigator, Charles Michalopoulos, Chief Economist, MDRC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018.01.415.00
Record Dates: First submitted 2014-02-26; First posted 2014-03-03 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Pregnancy; Postpartum Care; Infant Development
Keywords: Pregnancy; Postpartum programs; Infant health services
MeSH Terms: interventions — House Calls

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home visiting (Experimental): Home visiting group: Women will be randomized so that 60 percent can receive home visiting services and 40 percent are in the control group. Home visiting for low-income, pregnant women - whereby individualized in-home services (including direct education, assessments, and referrals to community resources) are provided to families - has been identified by the Strong Start initiative as one promising method for reaching women who are vulnerable to poor birth outcomes.
  Interventions: Behavioral: Home visiting
- Non-Home Visiting (No Intervention): Control group: As described above, women will be randomized so that 60 percent can receive home visiting services and 40 percent are in the control group.The home visiting program will provide control group families with referrals to other appropriate services in the community.

INTERVENTIONS:
Behavioral: Home visiting — MIHOPE-Strong Start will examine local programs that use either of two home visiting service models that have shown previous evidence of improving birth outcomes: Healthy Families America (HFA) and Nurse-Family Partnership (NFP). HFA and NFP provide disadvantaged expectant mothers with individualized in-home services, including assessment of prenatal and postnatal risks to child well-being; referrals to needed health care or social services; and direct education of parents by home visitors on such topics as healthy prenatal behaviors, parenting, and child development.
  Arms: Home visiting

SUMMARY:
Adverse birth outcomes result in significant emotional and economic costs for families and communities. Research suggests that poor birth outcomes are influenced by a variety of social, psychological, behavioral, environmental, and biological factors. Home visiting programs represent a promising means of impacting each of these areas.

The Mother and Infant Home Visiting Program Evaluation - Strong Start (MIHOPE-Strong Start) will evaluate the effectiveness of two evidence-based home visiting models at improving birth outcomes for women who are enrolled in Medicaid or CHIP. The two models to be studied - Healthy Families America (HFA) and Nurse-Family Partnership (NFP) - have both shown some evidence of improving birth outcomes in prior research.

The overall goals of the study are to determine whether home visiting programs improve birth outcomes and reduce health care costs in the child's first year. In addition, the evaluation is designed to investigate the features of local programs and of home visitation that lead to greater effects on birth outcomes and health care costs. The study includes an impact analysis to measure what difference home visiting programs make on maternal prenatal health and health care use, preterm birth and other birth outcomes, and infant health and health care use. It also includes an implementation analysis that will describe the families who participate and examine how the program models operate in their local and state contexts. The primary data used in the study are expected to be from surveys completed by families and home visiting staff, Medicaid and CHIP data, vital records, and program service records. Among families who are eligible for the study, random assignment will be used to select families for enrollment in home visiting services. Those selected for home visiting services will form the program group, and those not selected will form a comparison group. The research team will monitor both groups over time to see if differences emerge in the outcome areas mentioned above. Although the study will affect which families can enroll in home visiting services, no fewer families will be served as a result of the study.

DETAILED DESCRIPTION:
The study's conceptual framework has three broad aspects: (1) inputs (factors influencing service delivery), (2) outputs (services delivered) and (3) outcomes for families. Each site in MIHOPE-Strong Start will use either the NFP or HFA home visiting model.

Community resources provide a foundation from which programs operate and are considered an input that influence how services are provided to families. In particular, these determine the outside referral services available to home visiting programs and the opportunities available to families in both the program and control groups. By connecting pregnant women with services, home visiting programs can change mothers' health care use, health behaviors, and health status, which in turn can lead to improvements in birth outcomes. In communities where services are limited, however, home visiting programs may have limited capacity to improve mothers' connections to such supports. Furthermore, a program's ability to improve outcomes is influenced by the "treatment differential," or the difference between service receipt among families who receive home visiting and families who do not receive home visiting. The more that control group members receive services that are similar to those provided by HFA and NFP, the smaller the "treatment differential." Community context also includes community characteristics that could affect norms toward use of social services and health care, or other influences on control group help-seeking and program group responses to home visiting programs. These contextual factors can affect program impacts in both positive and negative directions. The service model defines the program plan. It includes information such as the intended goals of the home visiting program; the expected frequency, duration, and content of home visits; and intended linkages with other services.

The MIHOPE-Strong Start implementation study will document the extent to which the two evidence-based models and their local counterparts have defined clear, coherent, and well-specified service plans for helping parents to obtain prenatal care, other services needed to reduce the risk of poor birth outcomes, and infant health care in the first year of life - a critical prerequisite to delivering services that could affect these outcomes.

In MIHOPE-Strong Start, the "service model" can be defined at two levels: the service model is defined by the national evidence-based model and then it may be refined or adapted by the agency that is operating a local program. It is important to clearly understand how HFA and NFP define their models since these models showed efficacy in prior research. At the same time, local programs often deliberately adapt models to fit their local contexts. Given inconsistent impacts on birth outcomes in past studies, in fact, such adaptations could be one path to improvements in program impacts.

There are multiple organizational influences on how a home visiting program defines its service model and its implementation system. These organizations include the local program operator, the purveyor of the evidence-based model that has been adopted (HFA or NFP), the state MIECHV (Maternal, Infant, and Early Childhood Home Visiting Program) grantee (if the site is participating in MIECHV), and community organizations with which the local agency collaborates.

The implementation system includes the resources for carrying out the service model. It incorporates policies and procedures for staff recruitment, training, supervision and evaluation; assessment tools, protocols and curricula to guide service delivery; administrative supports; organizational climate regarding fidelity and the use of evidence-based practices; available consultation to address issues beyond the home visitor's skills and expertise; and the program's relationships with other organizations to facilitate referral and service coordination.

Other program characteristics that affect the services delivered include the attributes of staff in a given program. NFP specifies that home visitors should be registered nurses with a minimum of a baccalaureate degree in nursing. HFA gives local sites considerable discretion in this regard. Moreover, an individual staff person's own psychological well-being can influence how they approach their work with families. In addition to these global attributes, staff may vary in their degree of focus, confidence, and competence in carrying out responsibilities with respect to particular outcomes, due to variations in staff training and supervision. The implementation study will therefore be designed to understand the extent to which not only the service model, but also the implementation system and individual staff, are focused on activities that are expected to improve birth outcomes and maternal and infant health care use.

The attributes of families who enroll in a given home visiting program will also affect the program's opportunities to affect birth outcomes. HFA and NFP specify the characteristics of families that their programs can serve, yet even within each national model, local programs sometimes vary in the families they target either because of community characteristics, or because they vary in their processes for family recruitment. Baseline attributes of families who enroll can, in turn, influence services because staff are expected to tailor services to the family's strengths, needs, and concerns; because families vary in their understanding of the program and the benefits they are likely to derive from it; and because parents vary in their capacity, whether psychosocial or because of material resources, to engage with the services offered.

These inputs - the service model, implementation system, and characteristics of home visitors and families - all affect the outputs, or the services that families receive. Because home visiting programs rely heavily on referrals to other community organizations to meet families' needs, these outputs can include services provided directly by home visiting staff and referrals to other services.

NFP and HFA programs are designed to affect mothers' prenatal outcomes, including use of recommended levels of prenatal care, prenatal health behaviors related to birth outcomes such as smoking and use of alcohol or other substances, and mothers' prenatal health. These prenatal outcomes may influence birth outcomes, and birth outcomes may directly affect infant health outcomes, health care use and costs. By improving birth outcomes, parenting behaviors may also improve. Furthermore, home visiting services may indirectly improve infant health and health care use regardless of impacts on birth outcomes by improving parenting behaviors.

Based on this framework, MIHOPE-Strong Start will address the following broad research questions:

* What is the impact of home visiting programs that use one of these two evidence-based models on birth outcomes, maternal and infant health, and health care use up to the first year postpartum? How do impacts vary for key subgroups, such as smokers and young mothers?
* What is the impact of programs using each evidence-based model on the outcomes of MIHOPE Strong Start? The design is also intended to provide information that would allow actuaries at the Centers for Medicare and Medicaid Services (CMS) to estimate the effects of the programs on Medicaid costs.

The implementation study for MIHOPE-Strong Start will document the key features of HFA's and NFP's service models and implementation systems (at the national and local levels) that are expected to affect birth and health outcomes. The implementation research will answer these specific questions:

* How is each evidence-based service model - HFA and NFP - defined?
* How do local home visiting programs specify or adapt their service models relative to the national models with which they are affiliated?
* To what extent are local service models and implementation systems focused on preterm birth and related outcomes?
* What dosage of services do families actually receive in local programs and how much does it differ from the intended dosage?
* What kinds of referrals are provided to community services that could affect birth outcomes and the child's and mother's health?
* How do programs' inputs (such as the two evidence-based models, the extent of focus on birth outcomes, family characteristics, staff attributes, and community characteristics) relate to achieved outputs (in particular, the dosage of services received and referrals provided)?

Finally, the study will examine the intersection of impacts and implementation to answer the research question:

- How do home visiting programs using these two evidence-based models achieve their results?

To provide unbiased estimates of the effects of home visiting programs, families who are recruited into the study will be randomly assigned either to a program group that can receive home visiting services or to a control group that can use other services available in the community. Although the feasibility of carrying out random assignment must be assessed community-by-community, discussions with states and local programs thus far indicate that the need for home visiting services far exceeds the capacity of local programs in most places, allowing for the ethical creation of a control group. Other than home visiting services from the programs participating in MIHOPE-Strong Start, control group members can receive services available in the community for which they would normally be eligible. Control group members will receive referrals to such services. After their child reaches one year of age, those assigned to the control group will be able to receive home visiting services, if they are eligible for the local program. The evaluation will adhere to all ethical standards for program evaluation and has undergone human subjects review by the MDRC Institutional Review Board.

An impact analysis will estimate the effects of home visiting on prenatal health care use, birth outcomes, infant health, and maternal and infant health care use until the infant is one year old. The analysis will start with an analysis for the full sample, by evidence-based model (HFA and NFP), and for key subgroups. In all three cases, results will be presented for an "intent-to-treat" analysis that compares all program group members-regardless of whether they actually received home visiting services-with all control group members, some of whom may have received home visiting outside the MIECHV program. State Medicaid and vital records data will be collected from each of the 18 states and will provide all follow-up data, as well as some baseline data about sample members.

An implementation study, designed to complement the impact study, will collect information on community context, influential organizations, the service model, the implementation system, home visitors, families, and actual service delivery. The proposed evaluation will rely on multiple sources of data to understand how home visiting programs are implemented and what factors affect the quality of implementation. These data include information from each model's management information systems, interviews with home visitors and program managers at local sites, interviews with state administrators, and community characteristic information from the U.S. Census. Collecting basic implementation data across such a large number of sites will enable MIHOPE-Strong Start to provide evidence about which program variations are most effective at improving birth outcomes and maternal and infant health care use. It will also provide information about how programs can be designed to best improve these outcomes in the future.

ELIGIBILITY:
Inclusion Criteria:

* Must be pregnant with at least 8 weeks to expected due date
* Must be eligible for a home visiting program in MIHOPE-Strong Start
* Must be at least 15 years old

Exclusion Criteria:

* Currently enrolled in home visiting
* Does not speak English or Spanish

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1059 (Actual)
Dates: Start 2014-02; Primary Completion 2018-09 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Low birth weight | Time of birth
  Birth weight < 2,500 g
Preterm birth | Time of birth
  Birth at less than 37 weeks gestation
Infant admitted to the neonatal intensive care unit at birth | Time of birth
  Proportion of infants admitted to the NICU
Number of well-child visits for infant | During the first year of life
  Number of well-child visits during the first year of life, measured using Medicaid claims
Infant emergency department visits | During the first year of life
  Whether the infant was admitted to the emergency in the year after birth, measured from Medicaid claims data
Infant hospital admissions | During the first year of life
  Whether the infant was admitted to hospital in the year after birth, measured from Medicaid claims data
Any smoking during the 3rd trimester of pregnancy | Time of birth
  Whether the mother smoked during the 3rd trimester of pregnancy
Breastfeeding rates | Time of birth
  Infant was breastfed at hospital discharge, based on birth certificate data

SECONDARY OUTCOMES:
Fetal (intrauterine) growth | Time of birth
  By combining information on birth weight, gestational age, and the baby's sex, the prevalence of infants who are small for gestational age or large for gestational age will be estimated and examined.
Use of prenatal care | Time of birth
  Birth certificate data will be used to assess the date of the first prenatal care visit and the total number of prenatal care visits. In some states, particularly those with a low concentration of managed care, Medicaid data may also provide information to assess the effect of home visiting programs on prenatal care and the quality of data on prenatal care coming from birth certificates. These data, along with gestational age at birth, can be used to estimate the adequacy of prenatal care.
Emergency department use | During the first year of life
  From Medicaid files, number of infant visits to the emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Charles Michalopoulos, Ph.D., Study Director — MDRC; Virginia Knox, Ph.D., Study Director — MDRC; Keith Kranker, Ph.D., Principal Investigator — Mathematica Policy Research, Inc.; Anne Duggan, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- MDRC, New York, New York, United States

REFERENCES:
- [Background] Jill H. Filene, Emily K. Snell, Helen Lee, Virginia Knox, Charles Michalopoulos, and Anne Duggan (2013). The Mother and Infant Home Visiting Program Evaluation-Strong Start: First Annual Report. OPRE Report 2013-54. Washington, DC: Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.
- [Background] Lee, Helen, Anne Warren, Lakhpreet Gill (2015). Cheaper, Faster, Better: Are State Administrative Data the Answer? The Mother and Infant Home Visiting Program Evaluation-Strong Start Second Annual Report. OPRE Report 2015-09. Washington, DC: Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.
- [Background] Michalopoulos C, Lee H, Snell EK, Crowne S, Filene JH, Fox MK, Kranker K, Mijanovich T, Lakhpreet Gill L, and Duggan A. Design for the Mother and Infant Home Visiting Program Evaluation-Strong Start. OPRE Report 2015-63. Washington, DC: Office of Planning, Research and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.
- [Background] Lee, Helen, Sarah Crowne, Kristen Faucetta, and Rebecca Hughes. 2016. An Early Look at Families and Local Programs in the Mother and Infant Home Visiting Program Evaluation--Strong Start: Third Annual Report.
- [Background] Lee, Helen, Sarah Shea Crowne, Melanie Estarziau, Keith Kranker, Charles Michalopoulos, Anne Warren, Tod Mijanovich, Jill H. Filene, Anne Duggan, and Virginia Knox. (2019). The Effects of Home Visiting on Prenatal Health, Birth Outcomes, and Health Care Use in the First Year of Life: Final Implementation and Impact Findings from the Mother and Infant Home Visiting Program Evaluation-Strong Start. OPRE Report 2019-08. Washington, DC: Office of Planning, Research, and Evaluation, Administration for Children and Families, U.S. Department of Health and Human Services.
- See also: Link to the MIHOPE-Strong Start first annual report (cited above) — http://www.mdrc.org/sites/default/files/MIHOPE_SS_FR.pdf
- See also: MDRC's MIHOPE-Strong Start Project page — https://www.mdrc.org/project/mother-and-infant-home-visiting-program-evaluation-mihope-strong-start#featured_content
- See also: Link to the MIHOPE-Strong Start second annual report (cited above) — http://www.mdrc.org/publication/cheaper-faster-better-are-state-administrative-data-answer
- See also: Link to MIHOPE-Strong Start final report (cited above) — https://www.mdrc.org/publication/effects-home-visiting-prenatal-health-birth-outcomes-and-health-care-use-first-year-life